CLINICAL TRIAL: NCT06795282
Title: Effects of Three Different Root Canal Filling Materials Used in Single-Session Root Canal Treatment on Postoperative Pain: A Randomized Clinical Study
Brief Title: Post Operative Sensitivity of MTA Obturation
Status: Completed | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ayşe Tuğba Eminsoy Avcı, Principal Investigator, TC Erciyes University
Other Study IDs: AAvci
Record Dates: First submitted 2024-12-22; First posted 2025-01-28 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Dental Pulp Disease; Endodontically Treated Teeth; Endodontic Disease
Keywords: MTA; Post-op pain; Epoxy resin sealer; putty MTA
MeSH Terms: conditions — Dental Pulp Diseases; Tooth, Nonvital; Pain, Postoperative | interventions — Pemetrexed

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- powder-liquid MTA: The root canal will be filled with MTA at the end of the first session and patients will fill out a post-op pain form for 1 week.
  Interventions: Drug: MTA
- Putty MTA: The root canal will be filled with putty MTA at the end of the first session and patients will fill out a post-op pain form for 1 week.
  Interventions: Drug: MTA
- Epoxy resin sealer: The root canal will be filled with epoxy resin sealer and gutta-percha at the end of the first session and patients will fill out a post-op pain form for 1 week.

INTERVENTIONS:
Drug: MTA — MTA is primarily composed of tricalcium silicate, dicalcium silicate, bismuth oxide (for radiopacity), and small amounts of calcium sulfate. MTA is highly biocompatible, making it suitable for use in the root canal system and areas in close contact with tissues.
  Groups: Putty MTA; powder-liquid MTA

SUMMARY:
The aim of this study was to investigate the difference in postoperative pain caused by different root canal sealers in patients with irreversible pulpitis symptoms and no apical lesions.

ELIGIBILITY:
Inclusion Criteria:

* asymptomatic tooth with delayed positive response to thermal tests and electric pulp tests
* large pulp perforation during caries removal,
* inflamed pulp in which bleeding could not be controlled within 5 min,
* periodontally healthy mature mandibular first or second molar tooth.

Exclusion Criteria:

* patients if they were diabetic, immunocompromised, pregnant,
* had a positive history of antibiotic use during the past 1 month,
* required antibiotic prophylaxis
* used analgesic within 7 days prior to the beginning of treatment,
* were allergic to the materials used during root canal treatment,
* if the bleeding could be controlled within 5 min and vital pulp treatment could be performed,
* the tooth had negative response to vitality tests and/or was symptomatic,
* had an associated periapical lesion visible on a radiograph,
* needed a post-core or was planned to serve as prosthetic support,
* had a calcified root canal and internal or external root resorption,
* had tooth with open apex
* mandibular third molars

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Systemically healthy patients between the ages of 18-65
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
7-day postoperative pain after root canal treatment | 7 days
  At the end of the visit, patients were educated to record their postoperative pain level by assigning a number between 0 and 10 using the numerical rating scale (NRS) chart. They were categorized into four: 0=no pain, 1-3=mild pain, 4-6=moderate pain, and 7-10=severe pain. The patients were asked to record their pain level preoperatively, at 6, 12, and 24 h, and daily for up to 7 days, and return it to he investigators at a specific time.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University Faculty of Dentistry, Kayseri, Turkey (Türkiye)